CLINICAL TRIAL: NCT00651937
Title: Randomized Phase II Trial of Two Stem Cell Doses To Reduce Transplant Induced Symptom Burden in High Risk Patients With Multiple Myeloma or Amyloidosis
Brief Title: Trial of Two Stem Cell Doses To Reduce Transplant Induced Symptom Burden
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0601; NCI-2012-01687 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma; Primary Amyloidosis
Keywords: Multiple Myeloma; Primary Amyloidosis; Cytokine Modulation; Melphalan; Alkeran; Transplant Induced Symptoms; Stem Cell Infusion; Autologous stem cell transplant; ASCT; Granulocyte-colony stimulating factor; G-CSF; Apheresis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Melphalan; Surveys and Questionnaires; Granulocyte Colony-Stimulating Factor; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Dose (Active Comparator): Melphalan + Stem Cell Infusion (Standard Dose): Standard Dose (Arm 1) = Stem cell dose of between 4-6 x 10^6 cluster of differentiation 34 (CD34)/kg on Day 0. Melphalan 100 mg/m^2 via a Central Venous Catheter (CVC) Over 15-20 Minutes on Days -3 and -2 prior to stem cell infusion. Granulocyte-colony stimulating factor (G-CSF) 5 mcg/kg given subcutaneously (under the skin) on a daily basis for approximately 10 days. Beginning Visit 1, twice a week, paper and automated phone interview of symptoms and quality of life questionnaires.
  Interventions: Drug: Melphalan; Procedure: Stem Cell Infusion; Behavioral: Questionnaires; Drug: Granulocyte-colony stimulating factor (G-CSF); Procedure: Apheresis
- High Dose (Active Comparator): Melphalan + Stem Cell Infusion (High Dose): High Dose (Arm 2) = Stem cell dose of between 10-15 x 10^6 CD34/kg On Day 0. Melphalan 100 mg/m^2 via a Central Venous Catheter (CVC) Over 15-20 Minutes on Days -3 and -2 prior to stem cell infusion. Granulocyte-colony stimulating factor (G-CSF) 5 mcg/kg given subcutaneously (under the skin) on a daily basis for approximately 10 days. Beginning Visit 1, twice a week, paper and automated phone interview of symptoms and quality of life questionnaires.
  Interventions: Drug: Melphalan; Procedure: Stem Cell Infusion; Behavioral: Questionnaires; Drug: Granulocyte-colony stimulating factor (G-CSF); Procedure: Apheresis

INTERVENTIONS:
Drug: Melphalan — 100 mg/m^2 via a Central Venous Catheter (CVC) Over 15-20 Minutes on Days -3 and -2 prior to stem cell infusion.
  Other Names: Alkeran
Procedure: Stem Cell Infusion — Stem Cell Infusion is Day 0.
  Standard Dose (Arm 1) = Stem cell dose of between 4-6 x 10^6 CD34/kg On Day 0
  High Dose (Arm 2) = Stem cell dose of between 10-15 x 10^6 CD34/kg On Day 0.
  Other Names: Autologous Stem Cell Transplant; ASCT
Behavioral: Questionnaires — Beginning Visit 1, twice a week, paper and automated phone interview of symptoms and quality of life questionnaires.
  Other Names: Survey; Automated Phone Interview; M.D. Anderson Symptom Inventory; MDASI
Drug: Granulocyte-colony stimulating factor (G-CSF) — 5 mcg/kg given subcutaneously (under the skin) on a daily basis for approximately 10 days.
Procedure: Apheresis — Collection of stem cells from blood collected either through CVC or from a vein in one arm.

SUMMARY:
The goal of this clinical research study is to learn whether higher doses of stem cells can help to decrease the symptoms that occur after melphalan. Another goal of the study is to see how the dose of infused stem cells affects the levels of certain proteins in your blood. Researchers also want to learn how the dose of stem cells that you receive affects the quality of your life during the weeks after the transplant procedure.

DETAILED DESCRIPTION:
Stem cells are found in the bone marrow and bloodstream, and they rebuild blood, bone marrow, and the immune system. This study uses autologous stem cells, which are stem cells collected from your own blood. Melphalan is designed to damage the DNA (the genetic material) of cells, which may cause cancer cells to die. Granulocyte-colony stimulating factor (G-CSF) is designed to help the bone marrow to make more white blood cells. G-CSF is used in this study to help move your stem cells out of the bone marrow and into the bloodstream. If your doctor decides it is needed, you will also receive chemotherapy to help your blood stem cells move out of your bone marrow and into your blood. This allows the stems cells to be collected. Researchers also want to learn how the dose of infused stem cells affects the levels of certain cytokines in your blood. Cytokines are proteins that can cause symptoms such as fatigue and fever.

Treatment Plan:

If you are found to be eligible to take part in this study, you will need to have a central venous catheter (CVC) placed. A CVC is a flexible sterile tube that will be placed into a large vein that runs under your collarbone. Having the CVC allows blood to be drawn and medications to be given more easily and with less discomfort. You will be asked to sign a separate consent form to have the CVC placed, and the procedure will be more fully explained to you at that time.

If your doctor decides it is needed, you will receive chemotherapy to help your blood stem cells move out of your bone marrow and into your blood. You will be asked to sign a separate consent form for this chemotherapy.

Starting on the day of the stem cell infusion, you will receive G-CSF by injection under your skin. You will have the G-CSF injected once or twice a day for about 10 days. The injections may be given at home, if possible. You will be taught how to inject the G-CSF, or someone who agrees to be responsible for giving you the injections may also be taught.

Once the number of stem cells in your bloodstream is high enough, the stem cells will be collected over the course of 2-5 days. You will be asked to sign a separate consent form for the stem cell collection, and the process will be described in more detail at that time. Not counting the blood that is returned to you, about 32 tablespoons of blood will be drawn for the stem cell collection.

You will keep receiving the daily G-CSF injections on the days that your stem cells are collected. A procedure called apheresis will be used to collect the stem cells. During the apheresis, blood will be collected either through your CVC or from a vein in one arm. The blood will be processed through a machine to remove the stem cells, and then the rest of the blood will be returned to you through your CVC or through a vein in the other arm. The apheresis procedure will last several hours each time. You will be asked to sign a separate consent form for the apheresis procedure. You will have enough stem cells collected so that you will be able to have either 1 transplant with high doses of stem cells or 2 transplants with standard doses of stem cells. Your stem cells will be frozen (cryopreserved) until being given back to you.

About 2 weeks after your stem cells have been collected, you will have chemotherapy with melphalan. The melphalan will be given over 30 minutes through your CVC. Since this treatment destroys the normal bone marrow in addition to the myeloma cells, your blood stem cells must be given back to you. This is because blood stem cells are able to refill the bone marrow. If your doctor thinks it is needed, you may be admitted to the hospital the day before you receive melphalan to receive fluids by vein to hydrate you.

Two (2) days after receiving the melphalan, your previously collected stem cells will be unfrozen and given back to you through your CVC, similar to a blood transfusion. This is called an autologous stem cell transplant. You will be randomly assigned (as in the toss of a coin) to receive either a standard amount of stem cells or an experimental amount of stem cells. You have a 50/50 chance of being assigned to either group. After you receive your stem cells, you will be given G-CSF as an injection under the skin. You will keep having G-CSF injections until your white blood cell count returns to normal.

After your stem cells have been given back to you, it will take about 2 weeks for enough blood cells to be made. During this time, it is possible that you might not be making any blood cells. If this happens, you may need to have several red blood cell and platelet transfusions. You will receive antibiotics if infections occur, and you may need to be given feedings through the CVC.

The entire stem cell transplantation process will be done on an outpatient basis, if possible. Otherwise, you may need to stay in the hospital for up to 3-4 weeks.

After the stem cell transplant is completed, you will need to return to the clinic for follow-up visits at least once a week for a month, or more often if the doctor feels it is necessary. The follow-up visits will include the same tests and procedures as is standard of care. Research blood (about 2-4 teaspoons each time) will also be drawn on Day -2, Day 0, Day +3, Day +5, and Day +7; twice a week during weeks 2 and 3; and then once during week 4 for immune system tests.

Questionnaires and Physical Tests:

At several times during the study, you will be asked to complete a questionnaire about your symptoms and quality of life. Sometimes the questionnaire will be done over the phone with an automated phone system. Rating your symptoms using the telephone system should take less than 5 minutes for each call. The rest of the time questionnaires will be performed on paper and through phone interviews. You will also be asked to perform physical tests, including walking for 6 minutes and getting in and out of a chair.

The research nurse will teach you how to use the telephone system for measuring symptoms and your quality of life. You will perform the physical function tests and complete the symptom questionnaire. You will also have tests of the sensitivity of the nerves in your arms and legs. Blood (about 4-5 tablespoons) will be drawn for routine tests. Completing the questionnaires and tasks at this first visit should take about an hour.

During your hospital stay or clinic visits for the stem cell transplant, you will be asked on Day -2 (2 days before the transplant), Day 0, Day +3, Day +5, and Day +7 after the transplant to fill out a paper questionnaire that measures symptoms. You will also be asked on the same days to complete brief tasks that measure physical function.

During Weeks 2 and 3 you will be asked to fill out the paper questionnaire twice a week and complete the tasks of physical function once a week. During Week 4, you will be asked to fill out the questionnaire once and complete the tasks of physical function once. During Week 4, the sensory testing of the nerves in your arms and legs will also be repeated. On the same day as the physical tests, the research nurse will ask you to practice using the telephone system for measuring symptoms.

After you leave the hospital or clinic, the telephone system will call you at home. The calls will occur 1 time a week from Week 5 through Week 12 after the transplant, then 1 time a month during Months 3, 6, and 12 (+/- 1 month). The telephone system will ask you to rate how strong and tolerable the symptoms are, and how much the symptoms interfere with your daily life.

During the clinic visit that occurs about 90 days after the transplant, you will be asked to complete brief tasks that measure physical function, and you will also have the last test of the nerves in your arms and legs.

You will be on study for about 1 year.

This is an investigational study. Melphalan with autologous stem cell transplantation is FDA-approved for the treatment of myeloma and amyloidosis. The medications and treatment for this study are all commercially available. Up to 100 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma over the age of 60 in any of the following disease categories: a) Primary refractory disease b) Consolidation of a first partial or complete remission. OR
2. Patients with primary amyloidosis.
3. Zubrod PS of <2 or Karnofsky >/= 70.
4. Left ventricular ejection fraction >/= 40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
5. Forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusion capacity of lung for carbon monoxide (DLCO) >/= 40%. No symptomatic pulmonary disease.
6. Serum bilirubin </= 2 X upper limit of normal, serum glutamate pyruvate transaminase (SGPT) </= 4 X upper limit of normal. No evidence of chronic active hepatitis or cirrhosis. No effusion or ascites >1L prior to drainage.
7. HIV-negative.
8. Patient is not pregnant.
9. Patient or guardian able to sign informed consent.
10. Have greater than or equal to 10 x 10 e 6 CD34+ cells per kg of autologous stem cells cryopreserved for stem cell transplantation, procured with 5 or fewer apheresis collections.

Exclusion Criteria:

1) Patients unable to perform MDASI assessments due to language or cultural barriers.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Shah, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 13, 2008 to June 5, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Standard Dose Stem Cell Group: Patients undergoing ASCT for MM who were ≥60 years old or had AL amyloidosis were randomized to receive either a standard (4-6×106 cells/kg) of CD34+ cells after melphalan 200 mg/m2.
- High Dose Stem Cell Group: Patients undergoing ASCT for MM who were ≥60 years old or had AL amyloidosis were randomized to receive high dose (10-15×106 cells/kg) of CD34+ cells after melphalan 200 mg/m2.
Period: Overall Study
Arm/Group | Standard Dose Stem Cell Group | High Dose Stem Cell Group
Started | 39 | 41
Completed | 35 | 40
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Stem Cell Group | High Dose Stem Cell Group | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 79] | 65 [37 to 75] | 65 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 26 | 29 | 55
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Symptom Severity Burden as Measured by MDASI Scores
Description: MD Anderson Symptom Inventory (MDASI) Scale regularly administered during the first year following transplantation. This instrument is brief, easily understood, and provides a measure of the intensities of cancer-related symptoms. Participants rate the intensity of physical, affective, and cognitive symptoms on 0 to 10 numeric scales from "not present" (score of 0) to "as bad as you can imagine" (score of 10). Participants also rate amount of interference with daily activities caused by symptoms on 0 to 10 numeric scales from "did not interfere" (Score of 0) to interfered completely (score of 10).
Time Frame: The first 7 days post-transplant.
Population: Intention to treat analysis, all treated participants. One participant in High Dose group did not complete adequate number of MDASI's for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Dose Stem Cell Group | High Dose Stem Cell Group
Number analyzed (Participants) | 39 | 41
score on a scale | 4.27 (2.372) | 4.26 (2.264)

2. Primary Outcome: Mean Symptom Severity Burden as Measured by MDASI Scores
Description: MD Anderson Symptom Inventory (MDASI) Scale regularly administered during the first year following transplantation. This instrument is brief, easily understood, and provides a measure of the intensities of cancer-related symptoms. Participants rate the intensity of physical, affective, and cognitive on 0 to 10 numeric scales from "not present" (score of 0) to "as bad as you can imagine" (score of 10). Participants also rate amount of interference with daily activities caused by symptoms on 0 to 10 numeric scales from "did not interfere" (Score of 0) to interfered completely (score of 10)
Time Frame: 28 day course of ASCT
Population: Intention to treat analysis, all treated participants. One participant in High Dose group did not complete adequate number of MDSAIs for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Dose Stem Cell Group | High Dose Stem Cell Group
Number analyzed (Participants) | 35 | 40
score on a scale | 228.4 (191.0) | 223.0 (94.0)

ADVERSE EVENTS:
Time Frame: Adverse event collection through the last day of active treatment day 0 (stem cell infusion) up to 30 days as outlined in the treatment plan.
Arm/Group | Standard Dose Stem Cell Group | High Dose Stem Cell Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/40
Other Adverse Events (participants affected / at risk) | 1/35 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Stem Cell Group (N=35) | High Dose Stem Cell Group (N=40)
Graft Failure (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Stem Cell Group (N=35) | High Dose Stem Cell Group (N=40)
Graft Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes